CLINICAL TRIAL: NCT03123991
Title: Applying the Spanish Version of the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Adolescents as a Universal School-based Anxiety and Depression Prevention Program: a Cluster Randomized Controlled-trial
Brief Title: Applying the Spanish Version of the UP-A as a Universal School-based Anxiety and Depression Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Collaborators: Spanish Ministry of Education, Culture and Sport (Unknown); Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13/03315
Record Dates: First submitted 2017-03-16; First posted 2017-04-21 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): UP-A adapted as a preventive intervention. Specifically, the Spanish version of The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A) adapted as a 9 sessions school-based preventive intervention. The intervention is delivered in nine weekly sessions (each session lasting around 55 minutes).
  Interventions: Behavioral: UP-A adapted as a preventive intervention
- Wait-list Control Group (Other): Same than experimental group (EG), after EG finishes. Specifically, classes in waitlist condition will be offered the same intervention than experimental group after EG finishes the three months follow-up.Before that, waitlist means that the classess work as usual with issues of mental health.
  Interventions: Behavioral: Same than experimental group (EG), after EG finishes

INTERVENTIONS:
Behavioral: UP-A adapted as a preventive intervention — The Spanish Version of the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A) adapted as a school-based anxiety and depression preventive intervention. The UP-A (Ehrenreich-May et al., 2016) is a transdiagnostic anxiety and depressive disorders treatment protocol that implement a set of core principles to address common factors underlying youth anxiety and depressive symptoms in an individual setting. Core modules of the UP-A include: (1) Building and Keeping Motivation; (2) Getting to Know Your Emotions and Behaviors; (3) Behavioral Activation; (4) Sensational Awareness; (5) Being Flexible In Your Thinking; (6) Awareness of Emotional Experiences; (7) Situational Emotion Exposures and (8) Keeping it Going - Maintaining Your Gains.
  Arms: Experimental Group
Behavioral: Same than experimental group (EG), after EG finishes — The Spanish Version of the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A) adapted as a school-based anxiety and depression preventive intervention. The UP-A (Ehrenreich-May et al., 2016) is a transdiagnostic anxiety and depressive disorders treatment protocol that implement a set of core principles to address common factors underlying youth anxiety and depressive symptoms in an individual setting. Core modules of the UP-A include: (1) Building and Keeping Motivation; (2) Getting to Know Your Emotions and Behaviors; (3) Behavioral Activation; (4) Sensational Awareness; (5) Being Flexible In Your Thinking; (6) Awareness of Emotional Experiences; (7) Situational Emotion Exposures and (8) Keeping it Going - Maintaining Your Gains.
  Arms: Wait-list Control Group

SUMMARY:
The current study proposes to extend transdiagnostic treatment research to adolescents by establishing initial pre to post-treatment and follow-up outcomes associated with the use of the Spanish Version of the Unified Protocol for the Treatment of Emotional Disorders in Adolescents (UP-A; Ehrenreich-May, Bilek, Buzzella, Kennedy, Mash, & Bennett, 2016) as a universal school-based preventive intervention.

DETAILED DESCRIPTION:
The study has the primary aim to examine whether a transdiagnostic CBT intervention adapted as a school-based universal preventive intervention and delivered by professionals is more effective than the usual school curriculum in: (1) reducing symptoms of anxiety and depression and (2) preventing high levels of anxiety and depression from developing in 13-18 years old adolescents.

The study has the following secondary aims: (1) Examine the reduction in negative affect, anxiety sensitivity, emotional avoidance and emotional symptoms' interference levels at post-treatment as compared to pre-treatment levels; (3) Examine the improvement in positive affect, self-esteem, satisfaction with life, quality of life, school adjustment, and general indiscipline at post-treatment as compared to pre-treatment levels; (4) Examine the moderating role of gender, age, social economic status, personality traits, conduct problems, hyperactivity/inattention, and peer problems on the effectiveness of the UP-A program; (5) Assess the moderating role of home practice, understanding of basic concepts of the program, number of sessions attended, practice of specific strategies and behavior during sessions (6) Examine if the effects at post-treatment are maintained at the 3 month follow up; (7) Assess the feasibility and acceptability of implementing UP-A in a group format and in a school setting.

ELIGIBILITY:
Inclusion Criteria:

* Providing written, informed consent (both the adolescent and at least one of the parents or legal tutors)
* Being able to understand, write and read Spanish

Exclusion Criteria:

* No other exclusion criteria because of being an universal prevention study

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 157 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in Revised Child Anxiety and Depression Scale-30 (RCADS-30) at pre, post intervention and at 3 months follow-up. | Up to 3 months
  RCADS-30 is a widely-used questionnaire of self-reported anxiety and depressive symptoms in children and adolescents. The scale is comprised of six subscales derived from DSM-IV criteria: social phobia (SOC), generalized anxiety disorder (GAD), obsessive-compulsive disorder (OCD), panic disorder (PD), separation anxiety disorder (SAD), and major depressive disorder (MDD). All subscales except for the MDD can be summed to creat a Total Anxiety Disorder Symptoms Score. Each item is scored from 0 (= Never) to 3 (= Always), with higher scores representing more severe symptoms.
Change in Depression Questionnaire for Children [Cuestionario de Depresión para Niños] (CDN) (Sandín, Chorot, & Valiente, 2016) at pre, post intervention and at 3 months follow-up. | Up to 3 months
  The CDN is a 16-item self-report questionnaire designed to assess symptoms of DSM-IV major depressive disorder and dysthymic disorder in children and adolescents. In this study, the two items targeting suicidal ideation were not included because of indications from the school principal and school counseler implicated in the study. The items are rated on a 3-point scale of frequency corresponding to Never or almost never (=0), Sometimes (=1), and Very often (2). The sum of all items provides an overall score with higher scores indicated more elevated depression symptoms.
Change in Anxiety Scale for Children [Escala de Ansiedad para Niños] (EAN) (Sandín et al., 2016) at pre, post intervention and at 3 months follow-up. | Up to 3 months
  This 10- item questionnaire targeted to children and adolescents assesses anxiety symptoms during the last few weeks. Participants are instructed to respond to how frequently they have felt or experienced general anxiety symptoms on a four point, Likert-type scale, ranging from 0 (= Never or almost never) to 3 (= A lot of the times or almost always). The sum of all items provides an overall score with higher scores indicating more elevated anxiety symptoms.

SECONDARY OUTCOMES:
Strenghts and Difficulties Questionnaire (SDQ) (Goodman, 1997). | One week before and one week after after experimental group receives intervention; three months after experimental group finishes intervention and one week after wait-list control group finishes intervention
  The Spanish version by García and colleagues was used (García et al., 2000).
Children Positive and Negative Affect Schedule [Escalas PANAS para niños] (PANASN) (Sandín, 2003). | One week before and one week after after experimental group receives intervention; three months after experimental group finishes intervention and one week after wait-list control group finishes intervention
  This questionnaire is a downward version for children and adolescents aged 7-17 years of the Positive and Negative Affect Schedule for adults (Watson, Clark, & Tellegen, 1988).
Childhood Anxiety Sensitivity Index (CASI) (Silverman, Fleisig, Rabian, & Peterson, 1991). | One week before and one week after after experimental group receives intervention; three months after experimental group finishes intervention and one week after wait-list control group finishes intervention
  The Spanish version by Sandín and Chorot was applied (Sandín & Chorot, 1997).
Emotional Avoidance Strategy Inventory for Adolescents (EASI-A) (Kennedy & Ehrenreich-May, 2016). | One week before and one week after after experimental group receives intervention; three months after experimental group finishes intervention and one week after wait-list control group finishes intervention
  This measure is an adaptation of an adult measure of emotional avoidance (Fairholme, Ehrenreich-May, Ellard, Boisseau, Farchione, Barlow, 2008). The scale was adapted and translated to Spanish for this study.
Depression and Anxiety Interference Scale for children [Escala de Interferencia de Depresión y Ansiedad en Niños] (EIDAN) (García-Escalera, Sandín, Chorot, & Valiente, 2017). | One week before and one week after after experimental group receives intervention; three months after experimental group finishes intervention and one week after wait-list control group finishes intervention
  This scale measuring Depression and Anxiety Interference was created for this study.
Rosenberg Self-Esteem Scale (RSES) (Rosenberg, 1965) | One week before and one week after after experimental group receives intervention; three months after experimental group finishes intervention and one week after wait-list control group finishes intervention
  The Spanish adaptation by Chorot y Navas (1995; en Sandín, 2008) was used.
Satisfacion With Life Scale for Children (SWLS-C) (Sandín, Chorot, & Valiente, 2015). | One week before and one week after after experimental group receives intervention; three months after experimental group finishes intervention and one week after wait-list control group finishes intervention
  This measure is an adaptation for children and adolescents of an adult measure of satisfaction with life (SWLS) (Diener, Emmons, Larsen, & Griffin, 1985).
Kidscreen-10 (KIDSCREEN Group, 2006) | One week before and one week after after experimental group receives intervention; three months after experimental group finishes intervention and one week after wait-list control group finishes intervention
  The Spanish official version by the KIDSCREEN Group was used to measure quality of life (KIDSCREEN Group, 2006)
Schoool Adjustment Brief Scale [Escala Breve de Ajuste escolar] (EBAE-10) (Moral, Sánchez-Sosa, & Villarreal, 2010). | One week before and one week after after experimental group receives intervention; three months after experimental group finishes intervention and one week after wait-list control group finishes intervention
General Indiscipline Scale [Escala de Indisciplina General] (IG) | One week before and one week after after experimental group receives intervention; three months after experimental group finishes intervention and one week after wait-list control group finishes intervention
  Adapted from Martín and colleagues' questionnaire (Martín, Pros, Busquets, & Muntada, 2012)
Socio-Demographic Information Questionnaire | One week before and one week after after experimental group receives intervention; three months after experimental group finishes intervention and one week after wait-list control group finishes intervention
End of Program Questionnaire | One week before and one week after after experimental group receives intervention; three months after experimental group finishes intervention and one week after wait-list control group finishes intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bonifacio Sandín, PhD, Principal Investigator — Universidad Nacional de Educación a Distancia (UNED)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia-Escalera J, Valiente RM, Sandin B, Ehrenreich-May J, Prieto A, Chorot P. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A) Adapted as a School-Based Anxiety and Depression Prevention Program: An Initial Cluster Randomized Wait-List-Controlled Trial. Behav Ther. 2020 May;51(3):461-473. doi: 10.1016/j.beth.2019.08.003. Epub 2019 Aug 14. PMID 32402261
- [Derived] Garcia-Escalera J, Valiente RM, Chorot P, Ehrenreich-May J, Kennedy SM, Sandin B. The Spanish Version of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A) Adapted as a School-Based Anxiety and Depression Prevention Program: Study Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2017 Aug 21;6(8):e149. doi: 10.2196/resprot.7934. PMID 28827212